CLINICAL TRIAL: NCT02691728
Title: A Phase 4, Open-Label Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 1 and 4 HCV Infection With Autoimmune Disease
Brief Title: Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 1 and 4 HCV Infection With Autoimmune Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peter J. Ruane, M.D., Inc. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN_US-337-1748
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): 12 Week treatment with LDV/SOF FDC
  Interventions: Drug: LDV/SOF FDC

INTERVENTIONS:
Drug: LDV/SOF FDC

SUMMARY:
This study is evaluating the safety and efficacy of a 12 week treatment LDV/SOF FDC in patients with Chronic GT1 or GT4 HCV infection and autoimmune disease

ELIGIBILITY:
Inclusion Criteria:

* Chronic GT1 or GT4 HCV Infection
* Diagnosed with autoimmune disease (rheumatoid arthritis, psoriatic arthritis, lupus, etc.) and is currently receiving treatment for the condition.

Exclusion Criteria:

* Infection with HIV or HBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
SVR12 (Sustained Virologic Response) | Sustained Virologic Response 12 Weeks after Treatment Completion

CONTACTS AND LOCATIONS:
Locations (1):
- Peter J. Ruane, MD, Inc., Los Angeles, California, United States